CLINICAL TRIAL: NCT04463017
Title: A Double-blind, Placebo-controlled, Phase I Study of the Safety and Pharmacokinetics of Single Ascending Doses of HU6 in Healthy Volunteers
Brief Title: Ascending Dose Study of HU6 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Rivus Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RIV-HU6-101
Record Dates: First submitted 2020-07-03; First posted 2020-07-09 (Actual); Last update posted 2021-05-04 (Actual); Status verified 2021-05

CONDITIONS: NASH - Nonalcoholic Steatohepatitis
Keywords: NASH
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Intervention Model Description: The study will be conducted in one phase: a single dose, dose escalation phase in up to 7 cohorts
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Active Treatment: HU6 (Active Comparator): Planned doses of HU6; N = 74
  Interventions: Drug: HU6
- Placebo Comparator (Placebo Comparator): Non-active study drug N = 14
  Interventions: Drug: HU6

INTERVENTIONS:
Drug: HU6 — HU6 is designed to reduce the steatosis, inflammation, fibrosis and hepatocyte injury in Noncirrhotic Nonalcoholic Steatohepatitis (NASH)

SUMMARY:
This is a single ascending dose trial in healthy volunteers. The study will be conducted in up to 7 cohorts. Upon review of the safety and PK data, it may be decided to expand the current cohort versus dose escalate to the next cohort. In addition, the sponsor may elect not to enroll all 7 cohorts based on safety and/or PK and/or PD data.

DETAILED DESCRIPTION:
This is a single ascending dose trial in healthy volunteers. The study will be conducted in up to 7 cohorts. Upon review of the safety and PK data, it may be decided to expand the current cohort versus dose escalate to the next cohort. In addition, the sponsor may elect not to enroll all 7 cohorts based on safety and/or PK and/or PD data.

Up to 74 subjects will be enrolled to allow for replacement subjects, if deemed necessary. Fewer subjects may be enrolled if not all cohorts are utilized due to identification of the MTD in an earlier cohort.

Double-blind dosing will occur in cohorts 1 through 7. In these cohorts, 6 subjects will receive HU6 and 2 will receive matching placebo.

ELIGIBILITY:
TARGET POPULATION:

INCLUSION:

Subjects must meet all the following inclusion criteria to be eligible:

1. Male or female between 18 and 45 years of age, inclusive, at time of informed consent.

   1. Female subjects of childbearing potential must be non-lactating, not pregnant as confirmed by a negative urine pregnancy test at Screening and admission to Clinical Research Unit, and using, and agree to continue using, an effective method of contraception for at least 4 weeks prior to first study drug administration until 30 days after the last dose of study drug.
   2. Female subjects of non-childbearing potential must be surgically sterile (e.g., hysterectomy, bilateral tubal ligation, oophorectomy) or post-menopausal (no menses for >1 year with follicle stimulating hormone >40 U/L at Screening)
   3. Female subjects of childbearing potential must not donate ova during the study and for at least 30 days after the last dose of study drug.
   4. Male subjects who have not had a vasectomy and/or Subjects who have had a vasectomy but have not had 2 post surgery negative tests for sperm must agree to use an acceptable method of contraception from time of first dose of study drug until 30 days after the last dose of the study drug, and to not donate sperm during the study and for at least 30 days after the last dose of study drug.
2. Healthy per investigator judgment as documented by medical history, physical examination, vital sign assessments, 12-lead ECG, clinical laboratory assessments, and general observations.

   1. At Screening, abnormalities or deviations outside the normal ranges for any clinical assessments that are considered clinically significant by the Investigator (laboratory tests, ECG, vital signs) may be repeated once at the discretion of the Investigator(s), and results that continue to be outside the normal ranges must be judged by the investigator to be not clinically significant and acceptable for study participation.
   2. On admission to Clinical Research Unit, alanine aminotransferase (ALT), aspartate aminotransferase (AST), total bilirubin, and thyroid values must be within the upper limits of the normal range. Subjects with isolated elevation of bilirubin and presumptive Gilbert's syndrome are permissible. All other laboratory test results that are outside the reference range on admission to CRU and judged by the investigator to be not clinically significant may optionally be repeated. Results that continue to be outside the reference range must be judged by the investigator to be not clinically significant and acceptable for study participation.
   3. Subject must demonstrate clinical euthyroidism as assessed by a thyroid profile utilizing TSH and Free T4 testing at screening.
3. Body mass index between 18.0 and 30.0 kg/m2, with a minimum body weight of 45 kg for females and 50 kg for males, inclusive. Additional inclusion criteria for the high BMI single dose cohort:

   a. Body mass index > 30.0 kg/m2, waist circumference > 41"
4. Understands the procedures and requirements of the study and provides written informed consent and authorization for protected health information disclosure.
5. Willing and able to comply with the requirements of the study protocol.

EXCLUSION:

Subjects presenting with any of the following will not qualify for entry into the study:

1. Current or past clinically significant history of cardiovascular, cerebrovascular, pulmonary, gastrointestinal, hematologic, renal, hepatic, immunologic, metabolic, urologic, neurologic, dermatologic, psychiatric, or other major disease, as determined by the investigator. History of cancer (except treated non-melanoma skin cancer) or history of chemotherapy use within 5 years prior to Screening.
2. Any surgical or medical condition or history that, in the opinion of the investigator, may potentially alter the absorption, metabolism, or excretion of study treatment, such as, but not limited to gastric bypass surgery or small bowel resections.
3. Contraindication to study drug or its excipients and/or history of allergic or anaphylactic reactions.
4. Resting heart rate <45 or >100 bpm; blood pressure < 90 or >140 systolic, or <50 or >100 diastolic.
5. On screening ECG and by history:

   1. A marked baseline prolongation of QT/QTcF interval (e.g., repeated demonstration of a QTc interval > 450 msec for males and >470 msec for females).
   2. A history of additional risk factors for Torsades de Pointes (TdP) (e.g., heart failure, hypokalemia, family history of Long QT Syndrome).
6. Taking any of the following prohibited medications:

   For non-obese cohorts:

   a. Any prescription medication (with the exception of all hormonal contraceptives and hormone replacement therapies (oral, injectable, transdermal or implanted)) or over the counter multi-vitamin supplement, including products with CBD or any non-prescription products (including herbal-containing preparations but excluding acetaminophen) within 14 days prior to admission to CRU.

   For obese cohort:

   a. Limited background prescription medications are permitted to manage complications of obesity, but any drug known to inhibit or induce cytochrome P450 (CYP) enzymes and/or P-glycoprotein including St. John's wort (Hypericum perforatum) within 14 days or 5 half-lives (whichever is longer) prior to admission to CRU, is prohibited. Also prohibited is the use of concomitant medications that prolong the QT/QTc interval identified in the https://crediblemeds.org/ website list category of 'Known Risk'.
7. History of significant drug abuse within one year prior to Screening or use of soft drugs (such as marijuana) within 3 months prior to the Screening visit or hard drugs (such as cocaine, phencyclidine [PCP], opioid derivatives including heroin, and amphetamine derivatives) within 1 year prior to screening.
8. History of regular alcohol consumption exceeding 14 drinks/week [1 drink = 5 ounces (150 mL) of wine or 12 ounces (360 mL) of beer or 1.5 ounces (45 mL) of hard liquor] within 6 months of Screening.
9. Positive urine drug or urine alcohol test at Screening or on admission to CRU.
10. Current nicotine use or vaping regularly more than 5 cigarettes or the equivalent per week.
11. Consumed any food or drink/beverage containing grapefruit or grapefruit juice, apple or orange juice, pomelo juice, star fruit, Seville or Moro (blood) orange products within 6 days before admission to CRU. Vegetables from the mustard green family (e.g., kale, broccoli, watercress, collard greens, kohlrabi, brussels sprouts, mustard), food containing poppy seeds (e.g., muffins, bagels, and cakes) must not be consumed within 24 hours before admission to CRU.
12. Positive test results of hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab), or human immunodeficiency virus (HIV1/2) antibody.
13. Diabetes reflected by a fasting plasma glucose level of ≥126 mg/dL and a reflex HbA1c of ≥6.5%.
14. Participation in another clinical trial at the time of screening or exposure to any investigational agent within 30 days or 5 half-lives prior to admission to CRU, whichever is longer.
15. Donation of plasma within 7 days prior to dosing. Donation or loss of blood (excluding volume drawn at screening) of 50 mL to 499 mL of blood within 30 days, or more than 499 mL within 56 days prior to the first dosing.
16. Received a tattoo or body piercing (including ear piercings) within 2 months prior to Day 1, and/or significant open wound that may result in risk of infection.
17. Having a condition that the investigator believes would interfere with his/her ability to provide written informed consent, comply with study instructions, or which might confound the interpretation of the study results or put the subject at undue risk. Subjects with a history of hypo- or hyperthyroidism, peripheral neuropathy, malignant hyperthermia or chronic recurrent rash that is considered clinically significant by the investigator are excluded.
18. Must not be claustrophobic or have a history of claustrophobia, or intolerance of closed or small spaces.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2020-08-12 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Assess the dose relationship of PK Parameter Cmax | 3 months
  Following completion of each cohort, bioanalytical analyses for HU6, PK will be performed and plasma PK parameters for Cmax analyzed
Assess the dose relationship of PK Parameter AUC | 3 months
  Following completion of each cohort, bioanalytical analyses for HU6, PK will be performed and plasma PK parameters for AUC analyzed

CONTACTS AND LOCATIONS:
Overall Officials: Mark Matson, MD, Principal Investigator — Prism Research Clinic
Locations (1):
- Prism Clinical Research, Saint Paul, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No